CLINICAL TRIAL: NCT00192478
Title: A Phase 1/2, Open-Label, Repeat-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of MEDI-524, a Humanized Enhanced Potency Monoclonal Antibody Against Respiratory Syncytial Virus (RSV), in Children at Risk for Serious RSV Disease
Brief Title: Open-Label, Dose-Escalation Study of 2 to 5 IM Doses of MEDI-524 at 3 mg/kg or 15 mg/kg; Children to be Followed for 90 Days After Their Last Dose of MEDI-524
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP104
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — motavizumab

ARMS (1):
- 1 (Active Comparator): MEDI-524
  Interventions: Biological: Medi-524

INTERVENTIONS:
Biological: Medi-524 — IM doses of MEDI-524 administered at 3 mg/kg or 15 mg/kg at 30 day intervals

SUMMARY:
MEDI-524 given for up to 5 doses at 3 and 15 mg/kg to high-risk children appeared to be safe and well tolerated.

DETAILED DESCRIPTION:
This study is designed to describe the safety, tolerability, immunogenicity, and pharmacokinetics of escalating, repeated IM injections (the intended route of administration for immunoprophylaxis) of MEDI-524, initially in children £6 months old with a history of prematurity (³32 to £35 weeks gestation, without BPD), one of the target populations of infants at high risk for serious RSV disease.

ELIGIBILITY:
Inclusion Criteria:

* All male or female children must have met all the following criteria:
* [Groups 1, 2, and 3] The child must have been born at ³32 to £35 weeks gestation and have been £6 months of age at the time of entry into the study (child must have been entered on or before their 6-month birthday) or [Group 3 only] The child must have been £24 months of age at the time of entry into the study (child must have been entered on or before their 24-month birthday) and diagnosed with BPD, with stable or decreasing doses of diuretics, steroids, or bronchodilators within the previous 6 months
* The child must have been in general good health at the time of entry
* The child's parent or legal guardian must have provided written informed consent; and
* The child must have been able to complete the follow-up visits through 90 days following last injection of MEDI-524
* Parent/legal guardian of patient must have had available telephone access

Exclusion Criteria:

* Children must have had none of the following:
* Hospitalization at the time of study entry (unless discharge was expected within 3 days after entry into the study)
* [All children in Groups 1 and 2; only children £6 months of age in Group 3] Birth hospitalization >6 weeks duration or [Only children >6 months of age in Group 3] Birth hospitalization >12 weeks duration
* Been receiving chronic oxygen therapy or mechanical ventilation at the time of study entry (including CPAP)
* [Groups 1 and 2 only] Diagnosis of BPD, defined as history of prematurity and associated chronic lung disease with oxygen requirement for >28 days
* Congenital heart disease (CHD) (Children with medically or surgically corrected [closed] patent ductus arteriosus and no other CHD may be enrolled)
* Evidence of infection with hepatitis A, B, or C virus
* Known renal impairment, hepatic dysfunction, chronic seizure disorder, or immunodeficiency or HIV infection
* Mother with known HIV infection
* Any of the following laboratory findings in blood obtained within 7 days prior to study entry: BUN or creatinine >1.5´ the upper limit of normal for age; AST (SGOT) or ALT (SGPT) >1.5´ the upper limit of normal for age; hemoglobin <9.5 gm/dL; white blood cell count <4,000 cells/mm3; platelet count <120,000 cells/mm3
* Acute illness or progressive clinical disorder
* Active infection, including acute RSV infection
* Previous reaction to IGIV, blood products, or other foreign proteins
* Have ever received palivizumab
* Received within the past 120 days or currently receiving immunoglobulin products (such as RSV-IGIV [RespiGamÒ], IVIG), or any investigational agents
* Currently participating in any investigational study
* Previously participated in any investigational study of RSV vaccines or monoclonal antibodies.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2004-02; Primary Completion 2006-05 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Describe the safety and tolerability of repeated IM doses of MEDI-524 administered at 3 mg/kg or 15 mg/kg at 30 day intervals in children at risk for serious RSV disease | 30 days after patient's final dose of study drug
Pharmacokinetics of MEDI-524 | · Serum concentrations at each data collection visit will be summarized

SECONDARY OUTCOMES:
Immunogenicity of MEDI-524 | · Serum ELISA binding activity at each data collection visit will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Losonsky, MD, Study Director — MedImmune LLC
Locations (3):
- Argentina (2):
  - Hospital General de Niños "Ricardo Gutierrez", Buenos Aires
  - Hospital Interzonal General de Agudos "Dr. Diego Paroissien, Buenos Aires
- Hospital Clinico Pontificia Universidad Catolica de Chile, Santiago, Chile